CLINICAL TRIAL: NCT01944943
Title: Phase II Study of Vismodegib in Patients With Refractory or Relapsed B-cell Lymphoma or Chronic Lymphocytic Leukemia
Acronym: VISMOLY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VISMOLY
Record Dates: First submitted 2013-02-22; First posted 2013-09-18 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Diffuse Large B-cell Lymphoma; Indolent Non-hodgkin Lymphoma; Primary Central Nervous System Lymphoma; Chronic Lymphocytic Leukemia
Keywords: refractory/relapsed; diffuse large B-cell lymphoma; indolent non-hodgkin lymphoma; Primary central nervous system lymphoma; chronic lymphocytic leukemia
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vismodegib (Experimental): Vismodegib 150 mg will be administrated orally at a dosage of 150 mg (1 capsule) once a day during 12 months.
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: Vismodegib — 150 mg (1 capsule) of Vismodegib per day orally in continue during 12 months
  Other Names: GDC-0449, ERIVEDGE®

SUMMARY:
The purpose of this study is to determine the efficacy of Vismodegib drug in treatment of patients with relapsed or refractory B-cell lymphoma or chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
This is a multicenter open-label phase II study.

Primary objective:

To evaluate the efficacy of vismodegib in patients with relapsed/refractory B-cell lymphoma and CLL as measured by the best overall response rate (ORR) during the treatment period.

Secondary objectives:

* To evaluate the tolerability and the safety of vismodegib in patients with relapsed/refractory B-cell lymphoma and CLL
* To evaluate the efficacy of vismodegib in patients with relapsed/refractory B-cell lymphoma and CLL by measuring the overall (OR) and complete response (CR) rate during the study period, the maximum tumor shrinkage, the duration of response, the progression-free survival (PFS) and the overall survival (OS).
* To examine the expression of GLI-1 and other Hedgehog (Hh) signalling components in the tumor specimens before and during treatment with vismodegib and corresponding efficacy in patients.

  44 patients will be included in the study equally distributed into 4 cohorts according to their histological subtype:
* Cohort 1: 11 patients with Diffuse large B-cell lymphomas (DLBCL)
* Cohort 2: 11 patients with "indolent" lymphomas (iNHL): Follicular (FL), mantle cell (MCL) and marginal zone lymphoma (MZL) lymphoplasmacytic lymphoma (LPL)/ Waldenstrom macroglobulinemia (WM), small lymphocytic lymphoma (SLL)
* Cohort 3: 11 patients with Primary central nervous system lymphomas (PCNSL)
* Cohort 4: 11 patients with Chronic lymphocytic leukemia (CLL).

After 28 days screening period (Baseline), each patient will be treated by Vismodegib 150 mg per os during for a maximum of 12 months until disease progression, unacceptable toxicities, patient consent withdrawal, death, reasons deemed by the treating physician or study termination by the Sponsor.

Tumour assessment (clinical examination, laboratory tests, abdominal and chest CT scan (for PCNSL only at baseline), +/- PET scan for DLBCL, +/- brain MRI and CSF examination and ophthalmic examination for PCNSL, +/- bone marrow examination (except for PCNSL) will be performed at baseline, and then every 2 months during the first 6 months of treatment, and every 3 months thereafter until disease progression or up to 6 months after study treatment stop.

Response to treatment will be assessed also by Pharmacodynamic study in tumor samples by immunohistochimic and qPCR analysis at baseline and after one month of treatment with vismodegib.

Pharmacokinetic studies (before and after 1 month of treatment) will also be performed.

After study treatment discontinuation, the patients will be followed up every 3 months until disease progression or up to 6 months (after 1 year treatement).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of B-cell lymphoma (DLBCL, MCL, FL, MZL, LPL/WM, SLL or PCNSL) or CLL (Matutes score ≥4) requiring treatment that is recurrent after at least one prior therapy for which no potentially curative therapy nor better treatment option is available. Specifically, the patient should have received all treatments considered to be standards of care, including stem cell transplantation (when appropriate, if patient eligible), and agents known to have significant clinical efficacy in their disease.Patient must be eligible for tumor biopsy. Biopsy at relapse is mandatory for all patients except for PCNSL (optional) and should provide enough tumor tissue for biological tests (paraffin-embedded and frozen or RNAlater-conserved tissue).
* Age 18 and older
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
* Signed inform consent
* Life expectancy ≥ 3 months
* Patients who have received up to a maximum of 4 lines of treatment (including radiotherapy)
* Patients must have recovered from all toxicities related to prior treatments to ≤ grade 1.
* Adequate Laboratory Parameters (unless abnormalities are related to underlying disease) within 28 days prior to signing informed consent, including:

  * Absolute neutrophil count (ANC) ≥ 1000/μL
  * Platelet ≥ 75,000/μL
  * Hemoglobin > 8.5 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (UNL)
  * Hepatic enzymes (AST, ALT) ≤ 3 x institutional ULN
* Measurable disease:

  * Cohort 1 and 2 (DLBCL and iNHL): Bi-dimensionally measurable disease at CT scan with at least 2cm in their longest diameter.
  * Cohort 3 (PCNSL): Measurable PCNSL on MRI with gadolinium enhancement (no minimal size) or, for intraocular lymphoma (IOL), measurable disease at fundoscopic examination with elevated level of IL10 (>10 pg/ml) in the acqueous humor.
  * Cohort 4 (CLL): Measurable disease assessable in the blood (lymphocytosis, cytopenia) and/or by imaging (bi-dimensionally measurable disease at CT scan with at least 2cm in their longest diameter)
* Patient must be able to take oral medication
* Females of childbearing potential (FCBP) must :

  * have a negative pregnancy test (serum or urine, sensitivity < or = 25IU HCG/L) within 96 hours prior to starting study drug administration.
  * Agree to use two reliable forms of contraception or to practice complete abstinence from heterosexual contact during whole treatment period and up to 7 months after discontinuation of study drug treatment
* Male patients must agree :

  * to use a condom with female of childbearing potential or to practice complete abstinence during whole treatment period and up to 7 months after discontinuation of study drug treatment.
  * To abstain from donating semen during whole treatment period and up to 7 months after discontinuation of study drug treatment
* For all patients receiving vismodegib (GDC-0449):

  * To agree to abstain from donating blood during the whole study and for at least 7 months after discontinuation of study drug treatment
  * To agree not to share the study medication with another person

Exclusion Criteria:

* Pregnant or breastfeeding lactating females.
* For CLL patients, clinically significant auto-immune cytopenia, Coombs-positive hemolytic anemia as judged by the treating physician
* Concomitant anti-tumor therapy (e.g., chemotherapy, corticosteroids, other targeted therapy, radiation therapy). Corticosteroids may be authorized for PCNSL only during maximum 3 weeks (before and/or at the beginning of treatment with vismodegib) at a maximum dose of 1mg/kg of prednisone or equivalent.
* Use of any standard or experimental anti-cancer drug therapy within 28 days prior to the study drug therapy (Day 1).
* Patients with severe renal failure (creatinine clearance < 30 ml/min according to Cockcroft & Gault formula) and/or undergoing dialysis.

Note: Patients with moderate renal insufficiency (i.e. creatinine clearance ≥ 30 ml/min) may be included.

* Uncontrolled and/or unstable concomitant disease such as infection requiring treatment with intravenous antibiotics.
* HIV positive serology
* Active hepatitis B or C
* History of other disease, metabolic dysfunction, physical examination, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the study results or to expose the patient to high risk from treatment complications.
* Patients unable to comply with the protocol requirements according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The best overall response rate(ORR) | 12 months
  ORR will be measured by the best overall response (complete response (CR), uncofirmed complete response (CRu) or partial response (PR)) recorded during whole treatment period from the baseline until the end of treatment.
  ORR will be assessed according to Cheson 1999 for DLBCL and iNHL, according to Abey 2005 (IPCG response criteria) for PCNSL and to Hallek 2008 (IWCLL response criteria) for CLL.

SECONDARY OUTCOMES:
Overall Response rate | 2, 4, 6, 9, and 12 months
  Overall response rate will be evaluated as ORR, CR, CRu, PR, stable disease (SD) and progressive disease (PD) after 2, 4, 6, 9, and 12 months of treatment and every 3 months for 6 months after treatment discontinuation, until disease progression.
Progression Free Survival (PFS) | Up to 3 year
  Progression-Free Survival will be measured from the date of inclusion to the date of first documented disease progression, relapse or death from any cause. Responding patients and patients who are lost to follow up will be censored at their last tumor assessment date.
Response Duration | Up to 3 year
  Duration of response will be measured from the time of attainment of first CR, CRu or PR to the date of first documented disease progression, relapse or death from any cause. Subjects with no documented progression after CR, CRu or PR will be censored at the last tumor assessment date.
Overall survival | Up to 3 year
  Overall survival will be measured from the date of inclusion to the date of death from any cause. Alive patients will be censored at their last date known to be alive.
Correlation between Hedgehog (Hh) signaling in the tumor and the efficacy of Vismodegib | At baseline and at 28 days (+/- 7 days)
  Hh signaling cascade will be evaluated in tumors at baseline and at the end of cycle 1 (at Day 28 +/- 7 days) in order to:
  * Study pharmacodynamic of the drug (extinction of Hh signaling under treatment with Vismodegib)
  * Search for correlation between Hh signaling and clinical response to Vismodegib
Safety endpoints | Up to 2 year
  Description of all adverse events (AEs), laboratory data, vital signs and ECOG performance status, performed by cycle/visit and for the entire study.
Overall Response rate | 12 months
  Overall response will also be assessed using the Cheson 2007 criteria in patients with DLBCL. Patient without response assessment (due to whatever reason) will be considered as non-responder.

CONTACTS AND LOCATIONS:
Overall Officials: Roch HOUOT, MD, Principal Investigator
Locations (10):
- France (10):
  - Hôpital Henri MONDOR, Créteil
  - CHU Dijon _ Hôpital d'Enfants, Dijon
  - CHRU de Lille _ Hôpital Huriez, Lille
  - CHU de Nantes _ Hôtel Dieu, Nantes
  - Hôpital Saint-Louis, Paris
  - CHU Haut Lévèque, Pessac
  - CH Lyon Sud, Pierre-Bénite
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Hôpital René Huguenin _ Institut Curie, Saint-Cloud